CLINICAL TRIAL: NCT01860521
Title: Programmed Intermittent Epidural Bolus Versus Continuous Epidural Infusion for Second Trimester Voluntary Termination of Pregnancy Analgesia: a Randomized Study.
Brief Title: Programmed Intermittent Epidural Bolus Versus Continuous Epidural Infusion for Termination of Pregnancy Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Umberto Leone Roberti Maggiore, Principal Investigator, Research Fellow., IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCUL 4022
Record Dates: First submitted 2013-05-13; First posted 2013-05-22 (Estimated); Results first posted 2013-10-28 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-08

CONDITIONS: Medical; Abortion, Fetus
Keywords: Termination of pregnancy; Second trimester; Programmed intermittent epidural bolus; Continuous epidural infusion; Epidural analgesia; Legally Induced Abortion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Programmed Intermittent Epidural Bolus (Active Comparator)
  Interventions: Procedure: Programmed Intermittent Epidural Bolus; Procedure: Procedure of interruption of pregnancy; Drug: Drug used for analgesia procedures; Device: Pump for programmed intermittent bolus.; Drug: Drug used for termination of pregnancy procedure.
- Continuous Epidural Infusion (Active Comparator)
  Interventions: Procedure: Continuous Epidural Infusion; Procedure: Procedure of interruption of pregnancy; Drug: Drug used for analgesia procedures; Device: Pump for continuous epidural infusion.; Drug: Drug used for termination of pregnancy procedure.

INTERVENTIONS:
Procedure: Programmed Intermittent Epidural Bolus — An initial epidural loading dose consisting of 0.0625% levobupivacaine 20 mL (Chirocaine®, Abbott, Chicago, USA) plus sufentanil 10 µg (Fentatienil®, Angelini, Rome, Italy) was followed by 0.0625% levobupivacaine with sufentanil 0.5 µg/mL, 10 mL every hour, starting 60 minutes after the administration of the initial epidural loading dose until expulsion of the fetus. If the patient still felt pain (VAPS score ≥ 30mm), despite the analgesia, additional manual incremental boluses of 5-mL levobupivacaine 0.125% until the VAPS score was < 30 mm were administered.
  Arms: Programmed Intermittent Epidural Bolus
Procedure: Continuous Epidural Infusion — An initial epidural loading dose consisting of 0.0625% levobupivacaine 20 mL (Chirocaine®, Abbott, Chicago, USA) plus sufentanil 10 µg (Fentatienil®, Angelini, Rome, Italy) was followed by 0.0625% levobupivacaine with sufentanil 0.5 µg/mL at a rate of 10 mL/h, starting 60 minutes after the administration of the initial epidural loading dose until expulsion of the fetus. If the patient still felt pain (VAPS score ≥ 30mm), despite the analgesia, additional manual incremental boluses of 5-mL levobupivacaine 0.125% until the VAPS score was < 30 mm were administered.
  Arms: Continuous Epidural Infusion
Procedure: Procedure of interruption of pregnancy — Patients were administered 1 mg of gemeprost pessaries (Cervidil®, Merck Serono SPA, Roma, Italy) in the posterior fornix of the vagina every 3 hours up to 5 doses. If the expulsion of the fetus did not occur, the therapeutic regimen was repeated after 24 hours from the initiation of the treatment. Induction-to-abortion time (hours) was considered the period of time comprised between the first gemeprost pessary administration and fetal expulsion. Failure of induction of abortion was defined as women undelivered after two completed cycles (48h).The evacuation of the uterus under general anesthesia was performed if ultrasonography showed retained productions of conception.
Drug: Drug used for analgesia procedures — Levobupivacaine (Chirocaine®, Abbott, Chicago, IL, USA) and sufentanil(Fentatienil®, Angelini, Rome, Italy) were administered in both study groups according to the regimen of each intervention arm (Programmed Intermittent Epidural Bolus Versus Continuous Epidural Infusion).
  Other Names: Levobupivacaine: Chirocaine®, Abbott, Chicago, IL, USA.; Sufentanil: Fentatienil®, Angelini, Rome, Italy.
Device: Pump for programmed intermittent bolus. — Pump administering programmed intermittent epidural bolus for the maintenance of analgesia was used.
  Other Names: Pump: Gemstar®; Hospira, Lake Forest, USA.
  Arms: Programmed Intermittent Epidural Bolus
Device: Pump for continuous epidural infusion. — Pump administering continuous epidural infusion for the maintenance of analgesia was used.
  Other Names: Pump: Gemstar®; Hospira, Lake Forest, USA.
  Arms: Continuous Epidural Infusion
Drug: Drug used for termination of pregnancy procedure. — Gemeprost pessaries.
  Other Names: Gemeprost pessaries: Cervidil®, Merck Serono SPA, Rome, Italy.

SUMMARY:
This study included women who underwent voluntary second trimester termination of pregnancy. Patients were randomized to programmed intermittent epidural anesthetic bolus or continuous epidural infusion for pain analgesia. In this randomized, double-blind study, the investigators assess the incidence of motor block (primary outcome), degree of satisfaction of the patients, total levobupivacaine and sufentanil consumption and adverse events (secondary outcomes) between the two study groups.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* pregnancy at second trimester
* willingness of voluntary interrupt the pregnancy
* comprehension of Italian Language
* baseline pain score ≥ 30 on a 100-mm visual analog pain scale (VAPS)

Exclusion Criteria:

* contraindication to epidural analgesia and to narcotics
* history of drug abuse or chronic use
* maternal disease (such as severe asthma, cardiac, liver or kidney disease)
* inability to comprehend or comply with the analgesia pain management procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simone Ferrero, PhD, Study Director — Universita degli Studi di Genova; Umberto Leone Roberti Maggiore, MD, Principal Investigator — Universita degli Studi di Genova
Locations (1):
- Department of Obstetrics and Gynecology, San Martino Hospital and National Institute for Cancer Research, University of Genoa, Genoa, Ligury, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 2011 - June 2013. University Hospital.
Groups:
- Continuous Epidural Infusion: Pump : Pump administering either programmed intermittent epidural bolus or continuous epidural infusion for the maintenance of analgesia was used.
  Continuous Epidural Infusion : An initial epidural loading dose consisting of 0.0625% levobupivacaine 20 mL (Chirocaine®, Abbott, Chicago, USA) plus sufentanil 10 µg (Fentatienil®, Angelini, Rome, Italy) was followed by 0.0625% levobupivacaine with sufentanil 0.5 µg/mL at a rate of 10 mL/h, starting 60 minutes after the administration of the initial epidural loading dose until expulsion of the fetus. If the patient still felt pain (VAPS score ≥ 30mm), despite the analgesia, additional manual incremental boluses of 5-mL levobupivacaine 0.125% until the VAPS score was < 30 mm were administered.
- Programmed Intermittent Epidural Bolus: Pump : Pump administering either programmed intermittent epidural bolus or continuous epidural infusion for the maintenance of analgesia was used.
  Programmed Intermittent Epidural Bolus : An initial epidural loading dose consisting of 0.0625% levobupivacaine 20 mL (Chirocaine®, Abbott, Chicago, USA) plus sufentanil 10 µg (Fentatienil®, Angelini, Rome, Italy) was followed by 0.0625% levobupivacaine with sufentanil 0.5 µg/mL, 10 mL every hour, starting 60 minutes after the administration of the initial epidural loading dose until expulsion of the fetus. If the patient still felt pain (VAPS score ≥ 30mm), despite the analgesia, additional manual incremental boluses of 5-mL levobupivacaine 0.125% until the VAPS score was < 30 mm were administered.
Period: Overall Study
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus
Started | 52 (September 2011) | 52 (September 2011)
Completed | 52 (June 2013) | 52 (June 2013)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 52 | 104
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33.3 (4.7) | 32.4 (5.3) | 32.8 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 52 | 104
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 52 | 52 | 104

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Motor Block
Description: The assessment of the degree of motor block was performed in the right and left lower extremities using the Breen modified Bromage score: 1 = complete block (unable to move feet or knees), 2 = almost complete block (able to move feet only), 3 = partial block (just able to move knees), 4 = detectable weakness of hip flexion while supine (between scores 3 and 5), 5 = no detectable weakness of hip flexion while supine (full flexion of knees), and 6 = able to stand and to perform partial knee bend. Patients with a Bromage score < 6 were considered to have motor block.
Time Frame: Assessed every hour from starting the analgesia procedure (up to 66 hours from starting of the procedure).
Measure: Number; unit: participants
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus
Number analyzed (Participants) | 52 | 52
participants | 24 | 3
Statistical Analysis 1: Comparison: Continuous Epidural Infusion vs Programmed Intermittent Epidural Bolus; Test type: Superiority or Other; p < 0.001, Chi-squared

2. Secondary Outcome: Degree of Satisfaction of the Patients With the Analgesia Procedure
Description: At discharge from the hospital, patients were requested to answer the following question "Taking into consideration the variations in pain symptoms, as well as the adverse events experienced, if any, how would you define the grade of satisfaction with your analgesic treatment?" The grade of satisfaction was assessed using a visual analog scale (VAS) where 0 corresponded to "completely unsatisfied" and 100 to "completely satisfied".
Time Frame: At discharge from the hospital (up to 72 hours from starting of the procedure).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus
Number analyzed (Participants) | 52 | 52
mm | 73.2 (19.6) | 84.4 (15.2)
Statistical Analysis 1: Comparison: Continuous Epidural Infusion vs Programmed Intermittent Epidural Bolus; Test type: Superiority or Other; p = 0.005, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Total Levobupivacaine Consumption
Time Frame: At the moment of fetal expulsion (up to 66 hours from starting of the procedure).
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus
Number analyzed (Participants) | 52 | 52
mg | 86.2 (27.0) | 75.5 (26.8)
Statistical Analysis 1: Comparison: Continuous Epidural Infusion vs Programmed Intermittent Epidural Bolus; Test type: Superiority or Other; p = 0.047, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Total Sufentanil Consumption.
Time Frame: During the whole analgesia procedure (assessed between the starting of the procedure until 66 hours).
Measure: Mean (Standard Deviation); unit: microg
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus
Number analyzed (Participants) | 52 | 52
microg | 69.0 (21.6) | 60.4 (21.5)
Statistical Analysis 1: Comparison: Continuous Epidural Infusion vs Programmed Intermittent Epidural Bolus; Test type: Superiority or Other; p = 0.047, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus
Serious Adverse Events (participants affected / at risk) | 3/52 | 3/52
Other Adverse Events (participants affected / at risk) | 33/52 | 21/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Continuous Epidural Infusion (N=52) | Programmed Intermittent Epidural Bolus (N=52)
Hemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 3
Uterine perforation (Pregnancy, puerperium and perinatal conditions) | 2/35 | 0/37
OTHER ADVERSE EVENTS (reported when occurring in more than 1.9% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Epidural Infusion (N=52) | Programmed Intermittent Epidural Bolus (N=52)
Nausea (Gastrointestinal disorders) | 18 | 7
Hypotension (General disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 3 | 1
Pruritus (General disorders) | 14 | 17
Shivering (General disorders) | 11 | 9
Sedation (General disorders) | 3 | 0
Respiratory depression (General disorders) | 2 | 0
Failure of induction (Pregnancy, puerperium and perinatal conditions) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No